CLINICAL TRIAL: NCT00024687
Title: Study of SS1(dsFv)-PE38 (SS1P) Anti-Mesothelin Immunotoxin in Advanced Malignancies: IV Infusion QOD x Six Doses
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Support withdrawn - Study continued by NCI - see record NCT00006981
Sponsor: INSYS Therapeutics Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS1PE-002
Record Dates: First submitted 2001-09-24; First posted 2001-09-25 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms
Keywords: SS1(dsFv)-PE38 Anti-Mesothelin Immunotoxin; advanced malignancy
MeSH Terms: conditions — Neoplasms | interventions — SS1(dsFv)PE38

INTERVENTIONS:
Drug: SS1(dsFv)-PE38 (SS1P) Anti-Mesothelin Immunotoxin

SUMMARY:
Although Neopharm has terminated its sponsorship of this study, it is continuing under the sponsorship of the NCI. Please contact Raffit Hassan, MD at 301-451-8742 for more information. Also see the related NCI study "Experimental Drug SS1(dsFv)-PE38 to Treat Cancer" (Study ID number 010011).

SS1(dsFv)-PE38 is an oncology drug product containing a bacteria toxin, fused to a high affinity, disulfide stabilized antibody. The fused protein retains cell killing activity, but binds only to cells expressing mesothelin. Tumors characterized by very high surface mesothelin expression include mesothelioma; epithelial carcinomas of ovary and peritoneum; and squamous cancers of cervix and upper aerodigestive tract, including esophagus, head, and neck cancers.

This is a dose-escalating study to determine the maximum tolerated dose (MTD) of intravenous SS1(dsFv)-PE38 administered once every other day for six doses. Dose escalation will proceed in cohorts of 3 until dose-limiting toxicity (DLT) is observed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicities and maximum tolerated dose (MTD) of six doses of SS1(dsFv)-PE38 QOD administered by intravenous infusion to patients with advanced malignancies.

II. Characterize the plasma pharmacokinetics of SS1(dsFv)-PE38 after intravenous infusion.

III. Determine toxicities attributable to subsequent courses of SS1(dsFv)-PE38.

IV. Evaluate the response of selected advanced malignancies to intravenous infusion of six doses of SS1(dsFv)-PE38 QOD administered at the MTD.

V. Determine the induction of antibody against SS1(dsFv)-PE38 and its relationship to pharmacokinetics.

PROTOCOL OUTLINE: To exclude immediate allergic hypersensitivity reaction, each patient will receive a test dose of SS1(dsFv)-PE38, and be observed for 30 minutes prior to receiving study dosing. Each treatment will be given by intravenous infusion over 30 minutes every other day. Hydration will be maintained. (Oral hydration may be adequate, but intravenous hydration may be used at the Investigator?s discretion.) Patients will be observed for at least 4 hours after infusion on Day 1 of each treatment course to exclude immediate allergic reaction. Treatment may be repeated for a maximum of two additional courses after 4 weeks if re-treatment criteria are met. At least three patients will be accrued at each dose level. Dose escalation within a patient will not be allowed.

PROJECTED ACCRUAL: Up to 30 patients

ELIGIBILITY:
-Disease Characteristics-

Histopathologic diagnosis of one of the following malignancies: ovarian carcinoma, all non-mucinous epithelial histologies, including primary peritoneal and fallopian tube carcinoma; malignant mesothelioma, except sarcomatous histology; squamous cell cancer of the lung; squamous cell cancer of the cervix; or squamous cell cancer of the head and neck.

Tissue block must be available for analysis. Tumor, initial or recurrent, must be positive (at least 30% of tumor cells) for mesothelin by immunohistochemistry.

Recurrent unresectable disease after appropriate definitive therapy.

At least 4 weeks elapsed since any prior therapy, with recovery from side effects. No concurrent anti-tumor treatment of any kind.

Measurable or evaluable tumor documented within 4 weeks prior to study entry.

-Patient Characteristics-

At least 18 years of age.

At least 12-week life expectancy.

Performance Status (ECOG) 0-2.

Adequate organ function, including: Absolute neutrophil count at least 1,500/mm3; Platelets at least 75,000/mm3; Creatinine, Calcium, and total Bilirubin less than or equal to the upper limit of normal; Liver enzymes AST and ALT less than or equal 2.5 x the upper limit of normal; Albumin at least 3.0 g/dL; Oxygen (O2) saturation more than 93% (room air).

Informed Consent signed in accordance with institutional criteria.

No known central nervous system (CNS) or spinal cord involvement by tumor.

No detectable antibody to SS1(dsFv)-PE38.

No concurrent antitumor therapy.

No cardiovascular condition NY Heart Association Grade II-IV, or any clinically-significant pericardial effusion.

No infection requiring parenteral antibiotics; no HIV infection; and no seropositivity for Hepatitis B and Hepatitis C.

Must not be pregnant or nursing. Females of child-bearing potential must use an effective method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Locations (1):
- NCI/NIH, Bethesda, Maryland, United States